CLINICAL TRIAL: NCT02201615
Title: The Effect of Perineal Massage in Childbirth: the Rate of Episiotomy Procedures, Perineal Tears and the Length of the Second Stage of Labour
Brief Title: The Effect of Perineal Massage in Childbirth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Gulbahtiyar DEMİREL, Assistant Professor, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SBF - 005; GD01MD2958058 (Registry Identifier: GD01MD2958058)
Record Dates: First submitted 2014-07-23; First posted 2014-07-28 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Obstetric Labor Complications
Keywords: Perineal Massage; Episiotomy; Perineal Laceration
MeSH Terms: conditions — Obstetric Labor Complications | interventions — Parturition

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (1):
- Perineal Massage & Control (Experimental): Perineal Massage every 30 min, a 10 min 4 times in the first stage of labour, 1 times in the second stage of labour.
  Control routine care procedure at the clinic.
  Interventions: Other: Perineal massage in childbirth

INTERVENTIONS:
Other: Perineal massage in childbirth

SUMMARY:
Objective To examine the effects of perineal massage applied during the action of birth on the frequency of episiotomy procedures, perineal tearing and the duration of the second stage of birth.

Methods The present study was a randomized controlled experimental. Women (284 women) were informed on the study and provided their written consent. 10-minute perineal massage with glycerine was applied to the women in the test group for 4 times during the first stage and 1 time in the second stage of birth. The women in the control group received the routine care procedure at the clinic.

Results According to the study findings, 31% of the women in the test group and 69.7% of the women in the control group were made subject to episiotomy (p<0.05). In the test and control group 9.2%, 2.4% of the women developed spontaneous perineal laceration (p>0.05). The average duration of the action of birth was 25.33 minutes in the test group and 28.18 minutes in the control group (p<0.05).

Conclusion The study results indicate that perineal massage applied during the action of birth decreased the rate of episiotomy procedure and shortened the duration of the second stage of birth.

ELIGIBILITY:
Inclusion Criteria:

* With no pregnancy-related complications diagnosed during pregnancy,
* No definitive indication for C-section,
* Satisfying the pregnancy week in terms of the fetal dimensions,
* At the 37th-42nd gestation week,
* Applying to have her first or second birth,
* With no systemic condition,
* With head presentation,
* At the latent phase of the first stage of birth with a dilatation under 4 cm and effacement below 50%,
* That have provided written consent specifying their voluntariness in participating in the study.

Exclusion Criteria:

* With pregnancy-related complications diagnosed during pregnancy,
* Definitive indication for C-section,
* No satisfying the pregnancy week in terms of the fetal dimensions,
* At the <37th- >42nd gestation week,
* With systemic condition,
* With no head presentation,
* At the latent phase of the first stage of birth with a dilatation above 4 cm
* No have provided written consent specifying their voluntariness in participating in the study.

Ages: 19 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 284 (Actual)
Dates: Start 2010-01; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Episiotomy procedures | until completed the second stage of labour, about from 30 min to 24 h

SECONDARY OUTCOMES:
Length of the second stage of labour | until completed the second stage of labour, about from 30 min to 24 h

CONTACTS AND LOCATIONS:
Locations (1):
- Cumhuriyet University, Sivas, Turkey (Türkiye)

REFERENCES:
- [Derived] Demirel G, Golbasi Z. Effect of perineal massage on the rate of episiotomy and perineal tearing. Int J Gynaecol Obstet. 2015 Nov;131(2):183-6. doi: 10.1016/j.ijgo.2015.04.048. Epub 2015 Jul 26. PMID 26410801